CLINICAL TRIAL: NCT03137810
Title: Placental Cord Drainage Versus no Placental Drainage in the Management of Third Stage of Labour: Randomized Controlled Trial
Brief Title: Placental Cord Drainage Versus no Placental Drainage in the Management of Third Stage of Labour
Acronym: PLCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Shafy El Shahawy, Principal invesigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Placental Cord Drainage versus
Record Dates: First submitted 2017-04-04; First posted 2017-05-03 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Obstetric Delivery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placental cord drainage (Experimental): In 90 women after vaginal delivery of the baby, the placental end of the cut umbilical cord 1st will be clamped for few seconds and then unclamped and left open to drain blood in a vessel until flow stoped. This will prevent the drained blood from getting mixed with blood lost in the 3rd stage.
  Interventions: Procedure: placental cord drainage
- Non placental cord drainage (Active Comparator): In 90 women after vaginal delivery of the baby placental end of the cut umbilical cord will be kept clamped.
  Interventions: Procedure: non placemtal cord drainage

INTERVENTIONS:
Procedure: placental cord drainage — In the study group a of total number of 90 women placental end of the cut umbilical cord 1st will be clamped for few seconds and then unclamped and left open to drain blood in a vessel until flow stoped. This will prevent the drained blood from getting mixed with blood lost in the 3rd stage.
  Blood loss in the third stage will be measured using a Kelly's pad which will be used during delivery and the blood lost will be collected in a clean metal bowl which will be kept at the tail end of Kelley's pad.
  Arms: placental cord drainage
Procedure: non placemtal cord drainage — In 90 women after vaginal delivery of the baby placental end of the cut umbilical cord will be kept clamped.
  Arms: Non placental cord drainage

SUMMARY:
The aim of this work is to compare the effectiveness of placental cord drainage with no drainage in reducing the duration and blood loss in 3rd stage of labour.

ELIGIBILITY:
Inclusion Criteria:

* Full term Uncomplicated singleton pregnancy Pregnancy with vertex presentation Patients expected to have spontaneous vaginal delivery

Exclusion Criteria:

* Over distended uterus(hydramnios.large fetus) Previous history of postpartum haemorrhage Known coagulation disorder Haemoglobin less than 8 g/dl Ante partum haemorrhage Multiple pregnancies Instrumental delivery

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-11-01 (Estimated); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
Duration of the third stage of labour | within 15 min of delivery of baby

SECONDARY OUTCOMES:
Amount of blood loss | FIRST 24 HOURS
retained placenta | 1ST HOUR OF DELIVERY
Manual removal of placenta | 1HOUR OF DELIVERY
Changes in maternal haematocrit (Hct) after birth | 1ST 24 HOURS
blood transfusion | 1ST 24 HOURS

CONTACTS AND LOCATIONS:
Overall Officials: Hassan A Bayoumy, MD, Study Chair — Ain Shams University; Amgad E Abou-Gamrah, MD, Study Director — Ain Shams University
Locations (1):
- Ain shams university maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided